CLINICAL TRIAL: NCT00044551
Title: An Open Phase II, Multi Center Trial of BAY 59-8862 in Patients With Aggressive, Refractory Non-Hodgkin's Lymphoma
Brief Title: Evaluation of Bay 59-8862 in Patients With Aggressive, Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100389
Record Dates: First submitted 2002-08-30; First posted 2002-09-04 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Taxane; Lymphoma; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — taxane; Cytotoxins; IDN 5109

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Taxane (Cytotoxic, BAY59-8862)

INTERVENTIONS:
Drug: Taxane (Cytotoxic, BAY59-8862) — Daily 1 h infusion every 3 weeks

SUMMARY:
Almost two-thirds of lymphoma cases are Non-Hodgkin's Lymphomas (NHL). NHL is a malignant process that affects lymphoid cells found both in the lymph nodes and extranodally. Incidence and mortality rates from NHL are highest in developed countries. While many patients with aggressive NHL are curable with initial anthracycline-containing regimens, the majority of patients will relapse or prove refractory to initial therapy. The prognosis of patients with disease recurrence following a multidrug regimen is also limited. The current protocol is designed to test the safety and efficacy of BAY 59-8862 in patients with Aggressive Refractory Non-Hodgkin's Lymphoma.

ELIGIBILITY:
Inclusion Criteria: - Measurable disease as defined by the presence of at least one measurable lesion - Failed at least one prior therapy or has achieved remission but has progressed or relapsed within 6 months of therapy - Life expectancy of at least 12 weeks - Adequate bone marrow, liver and kidney function Exclusion Criteria: - Excluded medical conditions like: pre-existing neuropathy, active heart diseases or ischemia, serious infections, HIV infection, chronic hepatitis B or C, seizures, hypersensitivity to taxanes, organ transplants, some previous cancers - Excluded therapies and medications, previous and concomitant such as: anticancer chemotherapy or immunotherapy during the study or within 4 weeks prior to study entry; more than two prior anticancer chemotherapy regimens; radiotherapy during study or within 4 weeks prior to study entry; bone marrow transplant - Others: pregnant or breast-feeding patients; both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial; substance abuse, medical, psychological or social conditions that may interfere with the patient's participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2002-02; Study Completion 2003-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (23):
- United States (13):
  - Miami Beach, Florida
  - Chicago, Illinois
  - Shreveport, Louisiana
  - New Brunswick, New Jersey
  - Brooklyn, New York
  - Manhasset, New York
  - Syracuse, New York
  - The Bronx, New York
  - Valhalla, New York
  - Cleveland, Ohio
  - Memphis, Tennessee
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Edmonton, Alberta, Canada
- France (3):
  - Paris
  - Pierre-Bénite
  - Vandœuvre-lès-Nancy
- Germany (2):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Berlin, State of Berlin
- Netherlands (2):
  - Amsterdam
  - Groene Hilledijk
- United Kingdom (2):
  - Cambridge, Cambridgeshire
  - Maidstone, Kent